CLINICAL TRIAL: NCT06373276
Title: The Effects of a Home-Based Fall Prevention Program on Community-Dwelling Elderly's Fall Risk Category
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dilshaad Basrai Vad (Other)
Responsible Party: Sponsor-Investigator, Dilshaad Basrai Vad, Primary Investigator, Metro Physical Therapy
Organization: Metro Physical Therapy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1511
Record Dates: First submitted 2022-08-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Fall Risk
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants in the multiplanar balance training home-based exercise and educational group (group A) will have a video, as well as written instructions, of the intervention and dosage, along with the five educational brochures loaded on their phone via the SAFE beta app. In the SAFE beta app, the participants will be prompted daily to click on the beta app to watch the demonstration of the interventional exercise. They are then prompted to begin their daily prescriptive intervention, which is a 7-day-a-week program for 12 weeks. Participants can view a video of the exercise intervention in real-time in order to "mirror" the exercises as they are completing the exercises.
Who Masked: Investigator
Masking Description: The primary investigator, who delivers the treatment, is blinded to to the performance outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance training (Experimental): multiplanar balance training exercise with education
  Interventions: Other: multiplanar balance training exercise with education
- control (Placebo Comparator): Education only
  Interventions: Behavioral: education only

INTERVENTIONS:
Other: multiplanar balance training exercise with education — 7 minute daily balance training exercises
  Arms: Balance training
Behavioral: education only — 5 educational broshures
  Arms: control

SUMMARY:
The primary goal of this dissertation study is to determine if a home-based multiplanar balance training program with electronic assistance, will be effective in reducing one's fall risk category.

Hypothesis: After 12 weeks, there will be a statistically significant decrease in the fall risk category for individuals in a home-based multiplanar balance training and educational program with electronic assistance as compared to no change in the fall risk category for individuals in an educational control group with electronic assistance Hypothesis: To determine if an individual's fear of falling is lower following a home-based multiplanar balance training and educational program, with electronic assistance as compared to no change in fear of falling following an educational control group with electronic assistance post-intervention.

Hypothesis: An individual's quality of life will improve following a home-based multiplanar balance training and educational program, with electronic assistance as compared to no change in the quality of life following an educational control group with electronic assistance post-intervention.

Hypothesis: Adherence and feasibility will be greater with a home-based multiplanar balance training program, with electronic assistance as compared to a control group with electronic assistance.

Hypothesis: There will be a statistically significant inverse relationship between an individual's fear of falling and their fall risk category.

ELIGIBILITY:
Inclusion Criteria:

Age of 65 years or older

* Able to transfer and walk independently at least 10 feet without an assistive device
* Living independently (defined as transferring independently and perform activities of daily life independently) in a home, or condo in the community
* Maintain a single legged stance greater than or equal to 2 seconds and less than or equal to 10 seconds bilaterally
* A Mini-Cog test (a tool that assesses signs for dementia) score of 3 or greater (appendix IV)
* Possession of an I-Phone less than 7 years old
* Able to start within 2 weeks of enrollment

Exclusion Criteria:

* • Unable to comprehend spoken English or communicate verbally in English

  * Diagnosis of a central neurological disease
  * Diagnosis of cognitive disease
  * Surgery or hospitalization within the last 6 months
  * Active cancer and/or undergoing current treatment
  * Current utilization of a trainer
  * Current utilization of a physical therapist for gait, balance, or lower extremity issues

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Timed up and Go Test measured in Seconds | 1 minute
  walk 10 feet, turn around and walk back to start position
3 stage balance test measured in seconds | 20 seconds
  tandem gait stance measured up to 10 seconds
30-second chair stand measured in repeitions | 40 seconds
  Stand up from chair, sit back down and repeat for 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Metro PT, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic information along with outcome measures will be shared with the dissertation team.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after the trial ends. The data will be available for 6 months